CLINICAL TRIAL: NCT02873377
Title: A Novel Worksite Smoking Cessation Intervention for Hispanic Construction Workers
Brief Title: Smoking Cessation in Hispanic Construction Workers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Lee, PhD, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140019; 1R21CA202993-01A1 (NIH)
Record Dates: First submitted 2016-07-28; First posted 2016-08-19 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Smoking Cessation
Keywords: Hispanics; Construction workers; Tobacco Quitline; Nicotine replacement therapy
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Chewing Gum; Nicotine; Counseling

STUDY DESIGN:
Intervention Model Description: Study arms will be conducted simultaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Care (Experimental): Interventions: Nicorette Gum/Nicoderm CQ, Behavioral Smoking Cessation Counseling & Smoking Quitline Referral. Participants in the "Enhanced Care" intervention arm will receive a single face-to-face behavioral counseling session delivered at the construction site lunch truck, two brief follow-up phone counseling calls, fax referral to the Florida tobacco quitline (QL), and provision of up to 8 weeks of free Nicotine Replacement Therapy (up to 6 weeks provided by the study and 2 weeks provided by the QL). Participants in will receive two follow-up phone assessments at 3-, and 6-months of enrollment.
  Interventions: Drug: Nicorette Gum; Drug: Nicoderm CQ; Other: Smoking Quitline Referral; Behavioral: Behavioral Smoking Cessation Counseling
- Standard Care (Active Comparator): Interventions: Nicorette Gum/Nicoderm CQ, Smoking Quitline Referral. The "Standard Care" group (NRT) will receive fax referral to the Florida QL and provision of up to 8 weeks of free Nicotine Replacement Therapy (up to 6 weeks provided by the study and 2 weeks provided by the QL). Participants will receive two follow-up phone assessments at 3-, and 6-months of enrollment.
  Interventions: Drug: Nicorette Gum; Drug: Nicoderm CQ; Other: Smoking Quitline Referral

INTERVENTIONS:
Drug: Nicorette Gum — GlaxoSmithKline Nicorette Gum (nicotine replacement therapy)
  Other Names: NRT
Drug: Nicoderm CQ — GlaxoSmithKline Nicoderm CQ (nicotine replacement therapy)
  Other Names: NRT
Other: Smoking Quitline Referral — Fax referral to the State smoking Quitline
  Other Names: Quitline
Behavioral: Behavioral Smoking Cessation Counseling — One time face-to-face smoking cessation counseling and follow-up phone call
  Other Names: Counseling
  Arms: Enhanced Care

SUMMARY:
Construction workers have the highest rate of smoking among all occupations, and are frequently exposed to a wide range of workplace hazards (e.g. toxins), which interact with smoking to increase their health risks. Minority construction workers, in particular, have higher smoking and lower cessation rates compared to other groups, and they generally show lower access and participation in cessation and health promotion services. The number of Hispanic workers employed in the construction industry in the US has tripled in the past decade to 2.6 million (23% of all construction workers). This study will develop, administer, and evaluate a novel smoking cessation program in a hard-to-reach and underserved population of Hispanic male construction workers using using pilot cluster randomized clinical trial (RCT) to test the developed intervention for feasibility and potential efficacy.

DETAILED DESCRIPTION:
A two-arm, cluster-randomized controlled trial will be conducted with up to 15 construction sites, selected from one Construction Company in south Florida. Cluster randomization is used with construction site chosen as the unit of allocation because it is most practical in this setting and minimizes the risk of spillover effects from the intervention to the control group. In conjunction with the site's safety manager, the investigators will recruit 9 adult Hispanic construction workers per site (126 total) who smoke ≥5 cigarettes/day in the last year. Participants in the enhanced care will receive one culturally adapted brief face-to-face behavioral counseling session developed in phase 1 and delivered at a lunch truck, two brief follow-up phone counseling calls, fax referral to the Florida quitline (QL), and provision of up to 6 weeks of free NRT. Participants in the standard care will receive fax referral to the Florida QL, and provision of up to 8 weeks of free NRT.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic
* Construction worker
* Have smoked ≥ 5 cigarettes/day in the past year.
* Have access to telephone
* Have no plans to move in the next six months
* Are interested in making a serious quit attempt in the next 30 days
* Have no contraindication to NRT (e.g., history of hypersensitivity to nicotine, recent (past month) myocardial infarction, any history of serious arrhythmias or unstable angina pectoris, chronic dermatological disorder (e.g., psoriasis)).

Exclusion Criteria:

* Inability to understand consent procedures
* Not Hispanic
* Not a construction worker
* Haven't smoked ≥ 5 cigarettes/day in the past year.
* No access to telephone
* Has plans to move in the next six months
* Not interested in making a serious quit attempt in the next 30 days
* Has a contraindication to NRT
* Has a generalized chronic dermatological disorder (e.g., psoriasis)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Lee, PhD, Principal Investigator — University of Miami; Taghrid Asfar, MD, Study Director — University of Miami
Locations (1):
- Clinical Research Building University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asfar T, Arheart KL, McClure LA, Ruano-Herreria EC, Dietz NA, Ward KD, Caban-Martinez AJ, Samano Martin Del Campo D, Lee DJ. Implementing a Novel Workplace Smoking Cessation Intervention Targeting Hispanic/Latino Construction Workers: A Pilot Cluster Randomized Trial. Health Educ Behav. 2021 Dec;48(6):795-804. doi: 10.1177/1090198120960395. Epub 2020 Oct 16. PMID 33063570
- [Derived] Asfar T, McClure LA, Arheart KL, Ruano-Herreria EC, Gilford CG Jr, Moore K, Dietz NA, Ward KD, Lee DJ, Caban-Martinez AJ. Integrating Worksite Smoking Cessation Services Into the Construction Sector: Opportunities and Challenges. Health Educ Behav. 2019 Dec;46(6):1024-1034. doi: 10.1177/1090198119866900. Epub 2019 Aug 19. PMID 31426671
- [Derived] Asfar T, Caban-Martinez AJ, McClure LA, Ruano-Herreria EC, Sierra D, Gilford Clark G Jr, Samano D, Dietz NA, Ward KD, Arheart KL, Lee DJ. A cluster randomized pilot trial of a tailored worksite smoking cessation intervention targeting Hispanic/Latino construction workers: Intervention development and research design. Contemp Clin Trials. 2018 Apr;67:47-55. doi: 10.1016/j.cct.2018.02.007. Epub 2018 Feb 14. PMID 29454141

RESULTS

PARTICIPANT FLOW:
Period: Period 1: Enrollment
Arm/Group | Enhanced Care | Standard Care
Started | 65 | 69
Completed | 65 | 69
Not Completed | 0 | 0
Period: Period Title 2: 3 Months Follow up
Arm/Group | Enhanced Care | Standard Care
Started | 65 | 69
Completed | 43 | 47
Not Completed | 22 | 22
Not completed — Lost to Follow-up | 22 | 22
Period: Period Title 3: 6 Months Follow up
Arm/Group | Enhanced Care | Standard Care
Started | 65 | 69
Completed | 50 | 46
Not Completed | 15 | 23
Not completed — Lost to Follow-up | 15 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Care | Standard Care | Total
Number analyzed (Participants) | 65 | 69 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (1.5) | 38.2 (1.4) | 39.5 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 65 | 69 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 69 | 134
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 6 | 10 | 16
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 58 | 57 | 115

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Abstinence Rates
Description: Prolonged abstinence is defined as no smoking, not even a puff, after a grace period of two weeks after quit date. This will be assessed in follow up questionnaire and confirmed with saliva cotinine level of <15 ng/ml.
Time Frame: 6-month
Measure: Number; unit: Percentage of participants
Arm/Group | Enhanced Care | Standard Care
Number analyzed (Participants) | 50 | 46
Percentage of participants | 36.00 | 30.43

2. Secondary Outcome: 7-day Point- Prevalence Prolonged Abstinence Rate
Description: Point prevalence abstinence rates is defined as self report of not smoking; in the past 7 days not even a puff) confirmed by saliva cotinine level of <15ng/ml.
Time Frame: 6-month
Measure: Number; unit: Percentage of participants
Arm/Group | Enhanced Care | Standard Care
Number analyzed (Participants) | 50 | 46
Percentage of participants | 36.00 | 30.43

3. Secondary Outcome: Enrollment Rate
Description: Enrollment rate will be reported as the percentage of participants that were eligible and randomized against the participants screened.
Time Frame: Baseline
Population: Number of workers screened
Measure: Number; unit: Percentage of participants
Groups:
- All Workers Available - Before Randomization: All workers on constructions screened for eligibility
Arm/Group | All Workers Available - Before Randomization
Number analyzed (Participants) | 156
Percentage of participants
  Eligible Participants | 85.9
  Randomized participants | 85.9

4. Secondary Outcome: Quitline Response Rate
Description: Quitline Response will be reported by the percentage of participants that contacted the Quitline, enrolled in the tobacco Quitline and the participants that completed at least 1 phone call from Tobacco Quitline.
Time Frame: 6-month
Measure: Number; unit: Percentage of participants
Arm/Group | Enhanced Care | Standard Care
Number analyzed (Participants) | 65 | 69
Percentage of participants
  Contacted by tobacco Quitline | 49.2 | 40.6
  Enrolled in tobacco Quitline | 29.23 | 23.19
  Completed at least 1 phone calls from tobacco QL | 23.08 | 11.59

5. Secondary Outcome: Follow-Up Rate
Description: Follow up rate will be reported as the percentage of participants that completed their follow up visit.
Time Frame: 3-month, 6-month
Measure: Number; unit: Percentage of participants
Arm/Group | Enhanced Care | Standard Care
Number analyzed (Participants) | 65 | 69
Percentage of participants
  3-month follow-up | 66.15 | 68.12
  6-month follow-up | 76.92 | 66.67

6. Secondary Outcome: Questionnaire Response Rate
Description: Questionnaire response rate will be reported by the percentage of participants that completed the initial and follow up questionnaire.
Time Frame: 6-month
Measure: Number; unit: Percentage of participants
Arm/Group | Enhanced Care | Standard Care
Number analyzed (Participants) | 65 | 69
Percentage of participants
  completed initial questionnaire | 93.85 | 88.41
  Completed follow-up questionnaire | 76.92 | 66.67

7. Secondary Outcome: Rate of Compliance to Intervention
Description: Rate of compliance to intervention is reported as the percentage of participants who self-reported following intervention components at follow-up.
Time Frame: 6-month
Measure: Number; unit: Percentage of participants
Arm/Group | Enhanced Care | Standard Care
Number analyzed (Participants) | 65 | 69
Percentage of participants
  Counseling session + 2 phone calls | 43.08 | 88.40
  6 weeks NRT | 93.85 | 88.41
  4 Quitline counseling sessions | 6.15 | 2.9
  2 weeks NRT from Quitline | 15.38 | 13.04

8. Secondary Outcome: Change in Number of Cigarettes Smoked
Description: For the participants that did not quit, the change in number of cigarettes smoked will be reported as the number of cigarettes smoked per day at the 6 months follow up visit minus the number of cigarettes smoked per day at baseline
Time Frame: Baseline, 6-month
Measure: Mean (Standard Deviation); unit: Cigarettes smoked per day
Arm/Group | Enhanced Care | Standard Care
Number analyzed (Participants) | 50 | 46
Cigarettes smoked per day | -13.5 (1.5) | -11.5 (1.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Enhanced Care | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/69
Other Adverse Events (participants affected / at risk) | 0/65 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02873377/Prot_SAP_000.pdf